CLINICAL TRIAL: NCT01905345
Title: Influence of Consecutive Strength- and Endurance Regimes on the Myonuclear Domain and Satellite Cell in the M. Vastus Lateralis of Old Healthy Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REGPOT
Record Dates: First submitted 2013-07-16; First posted 2013-07-23 (Estimated); Last update posted 2017-08-07 (Actual); Status verified 2017-08

CONDITIONS: Regeneration Potential of Healthy Old Men in Terms of Satellite Cell Activation

STUDY DESIGN:
Who Masked: Participant

ARMS (3):
- Endurance and Resistance Training (Experimental): Endurance and resistance exercise
  Interventions: Procedure: Training
- Resistance Training (Experimental): resistance exercise (12wk)
  Interventions: Procedure: Training
- Resistance and resistance Training (Experimental): resistance exercise (24 wk)
  Interventions: Procedure: Training

INTERVENTIONS:
Procedure: Training

SUMMARY:
Randomised training intervention.

Influence of consecutive training regime on the impact of the myonuclear domain and satellite cell

Sarcopenia

Despite that the muscle mass can be positively influenced by training, the loading with high weights and/or to the total exhaustion is for many old persons not possible.

Therefore we aim to enhance the myonuclei in the muscle fiber of old male subjects in a first phase by endurance training, in order to promote a more effective muscle growth in a second phase by resistance exercise.

ELIGIBILITY:
Inclusion criteria: -male

* no fever at the beginning and during the study
* between 60 years and 75 years
* non smokers
* no known cardiovascular and orthopaedic problems
* no cardiac pacemaker
* fulfilling the health criteria

Exclusion criteria: -female

* fever or cold at the beginning or during the study
* non MRI compatible metal implants
* under 60 years or over 75 years
* smoker
* cardiovascular or orthopaedic problems
* cardiac pacemaker
* not fulfilling the health criteria

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-08; Primary Completion 2015-12 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Difference in % from baseline in fibre type specific number of satellite cells, fibre type specific myonuclear domain [um^2], myonuclear number [%] in response to consecutive training regimes | participants will be followed for the duration of training period, an expected average of 7 months
  Difference in % from baseline in fibre type specific number of satellite cells, fibre type specific myonuclear domain [um^2], myonuclear number [%] in response to consecutive training regimes

CONTACTS AND LOCATIONS:
Overall Officials: Hans H Jung, Prof MD, Principal Investigator — University Hospital Zurich, Division of Neurology
Locations (1):
- University Hospital Zurich, Division of Neurology, Zurich, Canton of Zurich, Switzerland